CLINICAL TRIAL: NCT05897385
Title: Analgesic Effect of IntraPeritoneal LIGNOcaine in Gynaecological Open Surgery: A Double-blinded Randomised Placebo-controlled Trial (IP LIGNO Trial)
Brief Title: Analgesic Effect of IntraPeritoneal LIGNOcaine in Gynaecological Open Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.1
Record Dates: First submitted 2023-05-21; First posted 2023-06-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Gynecologic Disease; Local Anesthetic Systemic Toxicity
Keywords: Lignocaine; Postoperative pain; Analgesia; Surgery; Gynaecological
MeSH Terms: conditions — Pain, Postoperative; Genital Diseases, Female; Agnosia | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Active Comparator): Intraperitoneal lignocaine 200mg/20mls + epinephrine 1:200,000
  Interventions: Drug: Lignocaine
- Group P (Placebo Comparator): Intraperitoneal 20ml of 0.9% normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lignocaine — Intraperitoneal lignocaine 200mg/20mls + epinephrine 1:200,000
  Other Names: INJECSOL LIG2
  Arms: Group L
Drug: Normal Saline — Intraperitoneal 20ml of 0.9% normal saline
  Other Names: B. Braun 0.9% Sodium Chloride Inj. B.P
  Arms: Group P

SUMMARY:
The incidence of postoperative pain is highly prevalent among surgical patients. Inadequate postoperative pain control can slow the recovery and it increases the risk of postoperative complications, namely lung collapse and chronic pain. Although morphine is the one of the gold standard analgesia option for postoperative pain, it comes with many unwanted adverse effects, such as severe nausea and vomiting, low blood pressure and dizziness. Thus, multimodal analgesia regime, including local anaesthetic (lignocaine) is strongly advocated for postoperative analgesia.

The normal route of lignocaine is injected into vein for the properties of analgesia and anti-inflammatory. It exerts its effect via the systemic absorption of drugs to block the central neuronal pain transmission. In recent years, studies have demonstrated that instillation of lignocaine inside abdominal cavity can reduce internal organ pain by blocking free nerve ending inside abdomen with minimal systemic absorption of drug and lower complications of systemic toxicity of local anaesthesia as compared to the intravenous route of lignocaine.

Several RCTs showed the beneficial effect of intraperitoneal lignocaine for the reduction of postoperative visceral pain after laparoscopic surgery. However, gynaecological open surgery (cystectomy, hysterectomy) involves greater degree of manipulation and trauma on the internal organs with greater visceral pain, resulting in longer duration of hospitalisation and delayed functional mobility recovery. It is believed that the intraperitoneal lignocaine reduces inflammatory response after surgery and exert analgesia effect by blocking the neural signal transmission at site of tissue injury. Therefore, it is important to conduct this study to examine the analgesic effect of intraperitoneal lignocaine in women undergoing gynaecological open surgery.

DETAILED DESCRIPTION:
Postoperative pain impedes the progress of recovery and increases the risk of postoperative complications, namely lung atelectasis, incidence of desaturation, pulmonary dysfunction and chronic pain. Although opioid is the one of the gold standard analgesia for postoperative pain, it comes with many unwanted adverse effects, such as respiratory depression, hypotension and incidence of nausea and vomiting. Thus, multimodal analgesia regime, including local anaesthetic is strongly advocated for postoperative analgesia.

Lignocaine is a local anaesthetic agent, which has the properties of analgesia, anti-inflammatory and anti-arrhythmia effect via the blockade of sodium channel receptor in the spinal cord and dorsal root ganglia. The intravenous lignocaine exerts its effect via the systemic absorption of drugs to block the central neuronal transmission. In recent years, studies have demonstrated that intraperitoneal route of lignocaine can reduce visceral pain by inhibiting peritoneal free nerve ending and reduce peripheral neuronal hyper-excitatory of pain signal transmission. It is also believed that intraperitoneal lignocaine is associated with minimal systemic absorption of drug and lower incidence of systemic toxicity local anaesthesia as compared to the intravenous route of lignocaine.

Several randomised controlled trials (RCTs) showed the beneficial effect of intraperitoneal lignocaine for the reduction of postoperative visceral pain after laparoscopic surgery. However, gynaecological open surgery has greater degree of organ manipulation and tissue injury with greater visceral pain, resulting in longer duration of hospitalisation and delayed functional mobility recovery. It is believed that the intraperitoneal lignocaine reduces inflammatory response after surgery and exert analgesia effect by blocking the neural pain signal transmission at site of tissue injury. The dosage of intraperitoneal lignocaine used in the literature ranged from 200-400mg. The serum concentration of intraperitoneal lignocaine was measured, which was associated with a relatively safe serum concentration of lignocaine. Pharmacological studies have showed that the adjuvant dose of adrenaline reduced the systematic absorption of intraperitoneal lignocaine. Therefore, this study is designed to examine the analgesic effect of intraperitoneal lignocaine in gynaecological open surgery. The investigators hypothesised that intraperitoneal lignocaine reduces postoperative pain score at rest and movement in women undergoing gynaecological open surgery.

ELIGIBILITY:
Inclusion Criteria:

* all adult women (American Society of Anesthesiologists (ASA) who >18 years old and <60 years old
* gynaecological open surgery with midline or transverse laparotomy incision (below or above umbilicus)

Exclusion Criteria:

* laparoscopic surgery
* allergic to lignocaine
* history of cardiac, vascular or liver disease
* ASA 3-5 or
* body mass index <18/ or >40

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | 1-hour after surgery in the recovery bay
  At rest and movement (0- no pain, 10- most pain)
Postoperative pain score | 24-hour after surgery in the ward
  At rest and movement (0- no pain, 10- most pain)
Postoperative pain score | 48-hour after surgery in the ward
  At rest and movement (0- no pain, 10- most pain)

SECONDARY OUTCOMES:
Postoperative patient-controlled analgesia morphine consumption | 24-hour after surgery in the ward
  Measured in milligrams
Postoperative patient-controlled analgesia morphine consumption | 48-hour after surgery in the ward
  Measured in milligrams
Number of patients requiring rescue analgesia | Throughout in recovery bay after surgery, on average 2-hour after surgery
  Number of patients
Postoperative nausea and vomiting | Throughout in the recovery bay after surgery, on average 2-hour after surgery
  Number of patients
Adverse events of lignocaine | Throughout the study completion, on average of 48 hours
  Central nervous system or cardiovascular side effects- arrhythmias, dizziness or numbness

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, MBBS, Principal Investigator — University of Malaya; Ka Ting Ng, MBChB, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perniola A, Magnuson A, Axelsson K, Gupta A. Intraperitoneal local anesthetics have predominant local analgesic effect: a randomized, double-blind study. Anesthesiology. 2014 Aug;121(2):352-61. doi: 10.1097/ALN.0000000000000267. PMID 24758776
- [Result] Williamson KM, Cotton BR, Smith G. Intraperitoneal lignocaine for pain relief after total abdominal hysterectomy. Br J Anaesth. 1997 Jun;78(6):675-7. doi: 10.1093/bja/78.6.675. PMID 9215018
- [Result] Patel R, Carvalho JC, Downey K, Kanczuk M, Bernstein P, Siddiqui N. Intraperitoneal Instillation of Lidocaine Improves Postoperative Analgesia at Cesarean Delivery: A Randomized, Double-Blind, Placebo-Controlled Trial. Anesth Analg. 2017 Feb;124(2):554-559. doi: 10.1213/ANE.0000000000001799. PMID 27984226
- [Result] Elhakim M, Elkott M, Ali NM, Tahoun HM. Intraperitoneal lidocaine for postoperative pain after laparoscopy. Acta Anaesthesiol Scand. 2000 Mar;44(3):280-4. doi: 10.1034/j.1399-6576.2000.440310.x. PMID 10714840
- [Result] Rademaker BM, Kalkman CJ, Odoom JA, de Wit L, Ringers J. Intraperitoneal local anaesthetics after laparoscopic cholecystectomy: effects on postoperative pain, metabolic responses and lung function. Br J Anaesth. 1994 Mar;72(3):263-6. doi: 10.1093/bja/72.3.263. PMID 8130042
- [Result] Shahin AY, Osman AM. Intraperitoneal lidocaine instillation and postcesarean pain after parietal peritoneal closure: a randomized double blind placebo-controlled trial. Clin J Pain. 2010 Feb;26(2):121-7. doi: 10.1097/AJP.0b013e3181b99ddd. PMID 20090438